CLINICAL TRIAL: NCT04444661
Title: Effects of COVID-19 Induced Deconditioning After Long-term High Intensity Resistance Exercise in Older Men With Osteosarcopenia A Randomized Controlled Trial
Brief Title: Effects of COVID-19 Induced Deconditioning After Long-term High Intensity Resistance Exercise
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Friedrich-Alexander-Universität Erlangen-Nürnberg (Other)
Responsible Party: Sponsor
Other Study IDs: FrOST-FU
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Osteoporosis; Sarcopenia
MeSH Terms: conditions — Osteoporosis; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIT-resistance exercise: High Intensity Resistance Exercise
- Non exercising control: Control group that maintained life style and physical activity habits

SUMMARY:
Osteosarcopenia designates the simultaneous presence of sarcopenia and osteopenia; both chronic conditions of advanced age. Dynamic-resistance exercise (DRT) might be the most powerful agent to fight osteosarcopenia. Indeed, in the present FrOST study, we clearly determine the positive effect of slightly adapted 18 month high-intensity (HIT)-DRT on bone mineral density (BMD), sarcopenia and other health related parameters in osteosarcopenic men. However, after a short training break, COVID-19 induced lock down prevented a re-start of the HIT resistance exercise training in the FrOST cohort.

The aim of the present observational study is thus to determine the effects of 6 months of deconditioning on health related parameters under special regard of osteosarcopenia in this cohort of older men with osteosarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* participants of the FrOST study (NCT03453463)

Exclusion Criteria:

* medication and diseases with potential impact on study outcomes during the last 26 weeks.

Ages: 74 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Study Population: Participants of the FrOST study (men 72 years and older with osteosarcopenia)
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
SMI | Change from Baseline to 26 weeks
  Skeletal muscle mass index (appendicular skeletal muscle mass / body height; kg/m2) as determined by Dual Energy x-Ray Absorptiometry

SECONDARY OUTCOMES:
BMD-LS | Change from Baseline to 26 weeks
  Bone Mineral Density at the Lumbar Spine as determined by Dual Energy x-Ray Absorptiometry
BMD-hip | Change from Baseline to 26 weeks
  Bone Mineral Density at the total hip as determined by Dual Energy x-Ray Absorptiometry
Sarcopenia-Z-Score | Change from Baseline to 26 weeks
  Z-Score of parameters constituting the metabolic syndrome (i.e. SMI, hand-grip strength, gait velocity)
Fat infiltration thigh muscles | Change from Baseline to 26 weeks
  Intramuscular adipose tissue at the mid thigh as determined by Magnetic Resonance Imaging
Fat infiltration para-vertebral muscles | Change from Baseline to 26 weeks
  Intramuscular adipose tissue at the mid thigh as determined by Magnetic Resonance Imaging
Maximum hip-/leg extensor strength | Change from Baseline to 26 weeks
  Maximum hip-/leg extensor strength as determined by an isokinetic leg press
Metabolic Syndrome Z-Score | Change from Baseline to 26 weeks
  Metabolic Syndrome Z-Score based on the definition of the International Diabetes Federation including waist circumference, resting glucose, HDL-cholesterol, triglyzerides, mean arterial blood pressure)
Self rated physical performance | Change from Baseline to 26 weeks
  Late-Life Function and Disability Index of McAuley et al.

CONTACTS AND LOCATIONS:
Overall Officials: wolfgang Kemmler, PhD, Principal Investigator — Institute of Medical Physics, Friedrich-Alexander University Erlangen-Nürnberg
Locations (1):
- Institute of Medical Physics, Friedrich Alexander University Erlangen-Nürnberg, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study are available from the corresponding author, [WK], upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: no limitation

REFERENCES:
- [Background] Kemmler W, Kohl M, Frohlich M, Jakob F, Engelke K, von Stengel S, Schoene D. Effects of High-Intensity Resistance Training on Osteopenia and Sarcopenia Parameters in Older Men with Osteosarcopenia-One-Year Results of the Randomized Controlled Franconian Osteopenia and Sarcopenia Trial (FrOST). J Bone Miner Res. 2020 Sep;35(9):1634-1644. doi: 10.1002/jbmr.4027. Epub 2020 Apr 28. PMID 32270891
- [Background] Lichtenberg T, von Stengel S, Sieber C, Kemmler W. The Favorable Effects of a High-Intensity Resistance Training on Sarcopenia in Older Community-Dwelling Men with Osteosarcopenia: The Randomized Controlled FrOST Study. Clin Interv Aging. 2019 Dec 16;14:2173-2186. doi: 10.2147/CIA.S225618. eCollection 2019. PMID 31908428
- [Derived] Kemmler W, Kohl M, Frohlich M, Schoene D, von Stengel S. Detraining effects after 18 months of high intensity resistance training on osteosarcopenia in older men-Six-month follow-up of the randomized controlled Franconian Osteopenia and Sarcopenia Trial (FrOST). Bone. 2021 Jan;142:115772. doi: 10.1016/j.bone.2020.115772. Epub 2020 Nov 26. PMID 33249320